CLINICAL TRIAL: NCT06785129
Title: Mechanisms Underlying Endometriosis and Migraine Comorbidity
Brief Title: Endometriosis and Migraine
Acronym: EMC
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Hadas Nahman-Averbuch, Assistant professor, Washington University School of Medicine
Other Study IDs: 202405127
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Migraine; Endometriosis
Keywords: Migraine; endometriosis; hormones; pain
MeSH Terms: conditions — Migraine Disorders; Endometriosis; Pain | interventions — carboxypeptidase M

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- migraine: patients with migraine
  Interventions: Device: Thermal stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Conditioned pain modulation (CPM) response; Biological: Hormonal assessment
- Endometriosis: patients with endometriosis
  Interventions: Device: Thermal stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Conditioned pain modulation (CPM) response; Biological: Hormonal assessment
- migraine and endometriosis: patients with migraine and endometriosis
  Interventions: Device: Thermal stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Conditioned pain modulation (CPM) response; Biological: Hormonal assessment
- control: healthy participants with no migraine or endometriosis
  Interventions: Device: Thermal stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Conditioned pain modulation (CPM) response; Biological: Hormonal assessment

INTERVENTIONS:
Device: Thermal stimuli — The Thermal Sensory Analyzer (TSA-II or PATHWAY platform - Medoc, Ramat Yishai, Israel) will be used to safely deliver heat and cold stimuli. These devices can deliver relatively complex stimuli via computer control. All targeted stimulus temperatures will be less than 50°C, and participants will be free to remove their arm or leg at any time from the thermode. Noxious cold stimuli will also be delivered with a plastic water container or a water bath (FISHER, USA). Participants will be free to pull out of the water bath at any time
Device: Pressure stimuli — Pressure stimuli will be applied by using a handheld algometer (Wagner Instruments) or the Pressure Algometer (Medoc, Ramat Yishai, Israel). These devices have a round probe that allows quantifying the amount of pressure that is being applied. The Pressure Algometer allows a real-time visual feedback to control and monitor applied pressure rates. Pressure will be applied to the lower leg, volar forearm, or trapezius.
Behavioral: Pain ratings — Pain intensity and pain unpleasantness ratings will be assessed.
Behavioral: Conditioned pain modulation (CPM) response — The CPM paradigm assesses endogenous inhibitory pain modulation efficiency. CPM testing includes the application of a "test" stimulus without conditioning (control run, pressure pain thresholds) and a subsequent application of the same test stimulus together with a conditioning stimulus (conditioning run, a 60 second of foot immersion in cold water). The CPM response is the difference in the pressure pain thresholds between the control and the conditioning runs.
Biological: Hormonal assessment — Blood samples (approximately 2 tablespoons) and/or saliva and/or urine will be collected for analyses of sex hormone levels (e.g., prolactin, testosterone, estradiol).

SUMMARY:
This study aims to determine differences in experimental pain and sex hormone levels between patients with migraine, patients with endometriosis, patients with migraine and endometriosis, and healthy controls. Participants will complete surveys, experimental pain paradigms and collection of samples for hormone analyses.

DETAILED DESCRIPTION:
Participants will be recruited via the pain, headache and Ob/Gyn clinics, via Volunteers for Health, via other studies in the lab, study staff, and via EPIC. When potential participants are inquiring about studies with the Pain the Lifespan Lab, the study team will describe this study among the options. Potential participants might be identified via EPIC records using age, sex, diagnoses, notes, problem list, medications, and phone number.

A research staff member will contact a potential participant and provide a description of the project. Potentially eligible participants will be invited to participate in the study, which will be conducted at Washington University School of Medicine. Participants will also be provided with a written summary of or the consent form for the study. The consent will be signed electronically using Docusign e-consent process either remotely during a phone call or a video call (WUSTL Zoom) with a study staff or in person.

After confirming the inclusion criteria and signing the consent form, participants will complete a 2.5-3 hour study visit of psychophysical assessments of thermal and pressure stimuli. Participants will also complete various questionnaires including demographic, social, health, behavioral, and psychological questionnaires. For adolescents, a parent/legal guardian will be asked to assist in completing some of the health-related surveys (i.e., physical developmental survey, health survey, migraine history survey). Obstetric, gynecologic, fertility, surgical history, medications, and pain will be abstracted from the medical record and/or via health history interview. Blood, urine, and/or saliva samples will be collected for hormonal, immune, and/or genetic testing. Additional samples will be stored in a biobank for future hormonal, immune and/or genetic analyses. Participants will then complete follow-up surveys once monthly for up to 1 year after the study visit which will assess changes to their pain symptoms and treatments. All study procedures are optional, and participants can stop or not complete tests if they want.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosed endometriosis, migraine, or both endometriosis and migraine
2. Healthy control subjects with no history of chronic pain
3. Age 12-45
4. Assigned female sex at birth

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Presence of prolactinoma
3. Presence of psychiatric, neurological, endocrinological and/or developmental conditions and taking medications for these conditions
4. Current use of dopamine agonist or SSRI medications
5. For patients aged 12-17 not having a parent/legal guardian willing to sign the consent and answer surveys about their child's health

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: participants with migraine OR with endometriosis OR with migraine and endometriosis OR with no chronic pain condition
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Conditioned pain modulation (CPM) response | Baseline
  This psychophysical test examine the inhibitory pain modulation efficiency. In this test, pressure pain thresholds (measures by kilopascal) are assessed before and during immersion of the foot in cold water.
Sex Hormones | baseline
  prolactin levels

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Nahman-Averbuch, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared after the completion of the study and based on a request